# **Official Title:**

A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination with mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 years

NCT: NCT06038617

IRB Document Date: August 12, 2024



Consent to Participate in a Research Study A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination with mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 years.

### **CONCISE SUMMARY**

This is a research study. Taking part in research is voluntary.

This study will look at fever and other side effects during the week following vaccination with COVID-19 and other routine childhood vaccines in children aged 6 months to under 5 years old. What we learn from this study may help doctors better understand side effects and health outcomes in children after vaccines.

Children in this study will be randomly assigned (like flipping a coin) to one of two groups. If your child is assigned to Group 1 they will receive routine childhood vaccines and the COVID-19 vaccine on the same day at Visit 1. One to three weeks later, they will have a health education telehealth visit (Visit 2). They will not receive any additional vaccines at Visit 2. If your child is assigned to Group 2 they will receive routine childhood vaccinations and not the COVID-19 vaccine on Visit 1. One to three weeks later, they will come back to the clinic to get the COVID-19 vaccine and receive health education at Visit 2. You will be asked to record your child's temperature and other symptoms for 7 days after each visit. Your child will continue to be monitored and you will be contacted by phone again 3 months after Visit 1 for a follow up Visit 3.

COVID-19 vaccine is routinely recommended for young children. As with every vaccine, there are risks associated with the COVID-19 vaccine that are described in this document. Some risks could include: redness, swelling or pain where the vaccine was given, fever, body aches, headache, fatigue, fussiness or irritability, sleepiness, decreased appetite, vomiting or diarrhea. Side effects should go away within a few days.

The total amount of time to be in this study is about three and a half months.

If you are interested in learning more about this study for your child, please continue reading below.

We are asking you to allow your child to take part in a research study because they are 6 months to under 5 years old and your child's healthcare provider has recommended that they receive a COVID-19 vaccine and at least one other routine childhood vaccine. Research studies are voluntary and include only people who choose to take part. Please read this consent form closely and take your time making your decision. The study doctor or study staff will discuss this consent form with you and your child. Please ask them to explain any words or information that you do not understand. We encourage you to talk with your family and friends before you decide to allow your child to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below.

Please tell the study doctor or study staff if your child is taking part in another research study.

This research study is supported by the Centers for Disease Control and Prevention (CDC). The CDC will pay a portion of the salaries for Dr. Michael Smith, Dr. Emmanuel Walter, and their research team to conduct the study.



Consent to Participate in a Research Study A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination with mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 years.

## WHO WILL BE MY CHILD'S DOCTOR ON THIS STUDY?

If you decide to have your child participate, Dr. Smith will be your child's study doctor and he will be in contact with your child's regular health care provider throughout the time that your child is in the study and afterwards, if needed.

## WHY IS THIS STUDY BEING DONE?

The Centers for Disease Control and Prevention (CDC) recommends that children receive multiple vaccines at the same visit, including COVID-19 vaccine. Available information supports the safety of giving vaccines at the same visit. Some children get fevers after they get vaccines. Fever that occurs after getting vaccines often occurs on the day of and the first few days following the vaccines. Rarely, the fever that occurs after vaccines may cause seizures in children. We are doing this study to see if giving young children routine vaccines on the same day without the COVID-19 vaccine and then giving the COVID-19 vaccine about one to three weeks later will result in a similar frequency of fever compared with giving the COVID-19 and other vaccines on the same day. We will also evaluate other symptoms and the health of your child after vaccination.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

About 600 children will take part in this study, in total. Children will take part in the study at 4 different hospitals and medical facilities. Around 160 children will take part at Duke University Health System.

# WHAT IS INVOLVED IN THE STUDY?

If you allow your child to be in this study, you will be asked to sign and date this form. If you do not want your child to be in this study, you should not sign this form. In this case, your child will still receive their usual care, but not as a part of this study.

We will also review the eligibility criteria with you to make sure your child qualifies for the study. Your child may participate in this study if they are recommended to receive a dose of COVID-19 vaccine and at least one other routine childhood vaccine that is not a live vaccine.

If the study team decides your child is eligible to participate in this study, he/she will be randomly assigned (by chance, like flipping a coin) to one of the 2 groups below:

- Group 1: COVID-19 and other routine vaccines will be given on the same day (Visit 1). One to three weeks later, your child will have a health education visit (Visit 2). He/she will not receive any vaccine at Visit 2.
- Group 2: Routine childhood vaccinations except COVID-19 vaccine will be given on the same day (Visit 1). One to three weeks later, your child will come back to the clinic to get the COVID-19 vaccine (Visit 2).



The group your child will be assigned to will be determined purely by chance. The study doctor, members of the study team or parents cannot choose the group to which a child will be assigned. However, you and your study doctor or study team will know if your child is assigned to the group who receives their routine childhood vaccines and COVID-19 vaccine at the same time, or if your child is assigned to the group who receives the COVID-19 vaccine one to three weeks following the other routine childhood vaccines.

All vaccines your child receives during the study will be recorded in his/her medical record and the State's immunization registry.

At Visit 1, parents of all children who take part in this study will be given health education materials and an age-appropriate toothbrush. You will also receive a thermometer.

The study activities are described further in the following:

# **VISIT 1 (DAY 1) AND FOLLOW-UP CONTACT:**

The following will happen:

- You will be asked questions about your child's health
- The study staff will:
  - o Take your child's temperature
  - o Give you a temporal scan forehead artery thermometer, a toothbrush, and health education materials
  - A study staff member will provide paper memory aids for both Visit 1 and Visit 2
  - o If you elect, the study staff will send you an electronic memory aid for Visit 1 through email or text to record your child's temperature and other symptoms he/she may have at home. Regardless of your decision, you will receive paper memory aids for Visits 1 and 2 to use in case the electronic system is down.
- Your child will be randomly assigned (like flipping a coin) to either receive routine childhood vaccines and the COVID-19 vaccine on the same day (Visit 1), or receive routine childhood vaccines during Visit 1 and return back to the clinic one to three weeks later to get the COVID-19 vaccine.
- Your child will receive the vaccines and will wait for 15 minutes afterwards
- You will schedule your child's next study visit (Visit 2)

At this visit, we will also ask you about the best way for the study team to contact you, which includes either telephone, text messaging, or email. We will ask you to choose how you would like to return your child's information that you record on the memory aid to the study team. You may elect to report your child's information on a daily basis using email or text messaging. This way is preferred and will require fewer contacts with the study team if done correctly. If this is not possible for you, you may



return your child's paper memory aid at the next study visit (Visit 2). You will need to tell us if you elect to use the internet or the paper memory aid alone at this visit.

You will also be given a temporal scan forehead artery thermometer to take home and keep. The study staff will instruct you on how to use it to measure your child's temperature at home. Using the provided thermometer, we will ask you to measure your child's temperature every evening after 4pm or right before your child goes to bed. You should measure your child's temperature at approximately the same time each evening, starting the evening of the day he/she receives the vaccines and for the next 6 evenings (a total of 7 evenings). You should record your child's temperature on the paper or electronic memory aid. If at any time during the entire 7-day period your child feels warm or you are concerned your child has a fever, you should also take his/her temperature. If at any time your child has a temperature of 100.4°F or greater, you should retake your child's temperature approximately 20 minutes later and record the highest temperature that you measured.

In addition to recording fever information, the study staff will also instruct you on how to use the paper or electronic memory aid to record other symptoms that your child may have. They will also teach you how to record whether your child received fever or pain medicines or received any medical attention.

We will ask you not to give your child fever or pain reducing medicines ahead of time to prevent fever or pain. However, you may give your child fever or pain reducing medicine after their vaccines if they develop fever or pain. If your child were to develop a high fever (a temperature of 102.2°F or 39°C or greater) or have a seizure with a high fever you should contact your child's doctor and study doctor.

If you selected text or email to report your child's information, we will call, text, or e-mail you approximately 2 days after enrollment if we do not see your child's temperature information reported or if the temperature information does not seem correct. At that time, we will obtain your child's temperature information over the phone or by e-mail and review instructions for using the internet. Further, we will call or e-mail you in approximately 8 days if your child's information was not recorded via the internet. At that call we will obtain missing information.

If you selected the paper memory aid alone to report your child's information, we will call or email you approximately 2 days after enrollment and obtain your child's temperature information. We will review instructions for using the memory aid and remind you to bring the memory aid to Visit 2. If your child received the COVID vaccine at Visit 1, we will provide a postage-paid envelope to return your memory aid.

## VISIT 2 AND FOLLOW-UP CONTACT

The following will happen:

• If your child did NOT receive COVID-19 vaccine at Visit 1, you and your child will return for a clinic visit and the study staff will:

- o Review your child's information that you reported after Visit 1
- o Review your child's health history and current medications
- o Give the COVID-19 vaccine, and you will need to wait for 15 minutes after the vaccine
- o Provide a new memory aid to record your child's temperature and other symptoms he/she may have
- o Provide education regarding dental care for young children
- If your child DID receive COVID-19 vaccine at Visit 1, you and your child may return for a clinic visit or a telehealth visit. The study staff will:
  - o Review your child's information that you reported after Visit 1
  - o Review your child's health history and current medications
  - o Provide education regarding dental care for young children
  - o Confirm that you have the paper memory aid for Visit 2, or send you an electronic memory aid for Visit 2 through email or text to record your child's temperature and other symptoms he/she may have

Using the thermometer given to you by the study team, you will be asked to measure your child's temperature the evening of Visit 2, and each evening for the following week, the same as for Visit 1. About 7 days after you finish reporting your child's temperature and other symptoms, we will ask you to complete a survey about your beliefs and preferences about childhood vaccines. If you choose to report by internet, you will get the survey by email or by text message. Otherwise, we will give you paper surveys at Visit 1to take home with you. We will give you a postage-paid envelope to return your memory aid and survey.

You can choose to continue reporting information the same way you did after Visit 1, or you can choose to switch from internet to paper reporting or vice versa, if you prefer. At this visit, we will reconfirm the best way for the study team to contact you, which includes either telephone, email, or text messaging.

# **VISIT 3 (APPROXIMATELY DAY 91)**

The following will happen:

- Study staff will
  - o Review your child's heath history and current medications via a telephone call

### HOW LONG WILL MY CHILD BE IN THIS STUDY?

Your child will be in this study for about 3 months. You and your child can choose to stop taking part at any time without penalty or loss of any benefits to which your child is entitled. However, if you and your child would like to stop participating in the study, we encourage you to talk to your child's doctor first to make sure they receive all of their needed vaccines.

DUHS IRB IRB NUMBER: Pro00113014

IRB REFERENCE DATE: 08/12/2024 IRB EXPIRATION DATE: 09/06/2025



Consent to Participate in a Research Study A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination with mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 years.

## WHAT ARE THE RISKS OF THE STUDY?

As a result of your child's participation in this study, he/she is at risk for the following side effects. You should discuss these with the study doctor and your child's regular health care provider if you choose.

## **COVID-19 Vaccine Risks**

With every medicine, including vaccines, there is a chance of side effects. There may also be risks, discomforts, drug interaction or side effects from these vaccines that are not yet known. The potential side effects from these study vaccines will not be different from what your child would experience if you received these vaccines as part of your regular care.

Possible risks with receiving the COVID-19 vaccine include:

- Redness, swelling, or pain where the vaccine was given
- Fever, body aches, headache, or fatigue
- Fussiness or irritability
- Sleepiness
- Decreased appetite
- Vomiting or diarrhea

Other possible risks of COVID-19 vaccine are:

- Severe allergic reactions
- Non-severe allergic reactions such as rash, itching, hives, or swelling of the face
- Myocarditis (inflammation of the heart muscle)
- Pericarditis (inflammation of the lining outside the heart)

Some people feel faint or actually faint after having received a vaccine. As with any vaccine or medication, there is a very small chance of a serious allergic reaction although researchers do not expect this to occur.

There may be risks, discomforts, drug interactions, or side effects that are not yet known.

# **Delay of COVID-19 Vaccine**

There is a potential risk of a short delay in protection against COVID-19 by delaying the COVID-19 vaccine by one to three weeks. If your child develops COVID-19-like symptoms (such as fever, cough, sore throat, or headache), you should consult with their health care provider. Their health care provider may order tests to see if they have COVID-19.

ARE THERE BENEFITS TO TAKING PART IN THE STUDY?



If you agree to allow your child to take part in this study, there is no direct benefit to your child. Parents may learn from the health education they receive for their child. We hope that in the future that information learned from this study may benefit other children who receive childhood vaccines.

## WILL MY CHILD'S INFORMATION BE KEPT CONFIDENTIAL?

Participating in research involves some loss of privacy. We will do our best to make sure that information about your child is kept confidential, but we cannot guarantee total confidentiality. Your child's personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information in order to conduct the research. Your child's personal information may also be given out if required by law.

As part of the study, results of your child's study-related laboratory tests and procedures may be reported to the CDC and its affiliates. In addition, your child's records may be reviewed in order to meet federal or state regulations. Reviewers may include representatives from the CDC, the Duke University Health System Institutional Review Board, and others as appropriate. If any of these groups review your research record, they may also need to review your entire medical record.

The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your and your child's privacy. With this Certificate, the investigators may not disclose research information that may identify you or your child in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use. Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:

- 1) there is a law that requires disclosure, such as to report child abuse or communicable diseases but not for legal proceedings.
- 2) you have consented to the disclosure, including for your medical treatment; or
- 3) the research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project or for information that is required by the Food and Drug Administration (FDA).

You should understand that a Confidentiality Certificate does not prevent you, your child, or a member of your family from voluntarily releasing information about your child's involvement in this research. If you want your child's research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy.

Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.



## WHAT WILL HAPPEN TO MY CHILD'S STUDY INFORMATION?

The study results will be retained in your child's research record until your child reaches the age of 21 years. At that time either the research information not already in your child's medical record may be destroyed or information identifying your child will be removed from such study results at Duke University Health System. Any research information in your child's medical record will be kept indefinitely.

Some information collected in research studies is maintained in your child's medical record. However, for this study that information will be inaccessible until the end of the study, unless your physician(s) decide that it is necessary for your child's care.

Your child's data may be stored and shared for future research without additional informed consent if identifiable private information, such as your child's name and medical record number, are removed. If your child's identifying information is removed from their data, we will no longer be able to identify and destroy them.

The use of your child's data may result in commercial profit. You and your child will not be compensated for the use of the data other than what is described in this consent form.

Some information collected in research studies is maintained in your child's medical record. However, for this study some information will be inaccessible until the end of the study, unless your child's physician(s) decide that it is necessary for your child's care.

This information may be further disclosed by the sponsor of this study. If disclosed by the sponsor, the information is no longer covered by federal privacy regulations. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your child's name or other personal information will not be revealed.

Some people or groups who receive your child's health information might not have to follow the same privacy rules. Once your child's information is shared outside of the Duke University Health System, we cannot guarantee that it will remain private. If you decide to share your child's private information with anyone not involved in the study, the federal law designed to protect your child's health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

## WHAT ARE THE COSTS TO YOU?

There are no costs to you or your child for being in this this study. However, routine medical care (care your child would have received anyway) will be charged to you or your child's insurance company. You may wish to contact your insurance company to discuss this further. In order to make sure that tests and



studies done solely for research purposes are not charged to you, we will carefully monitor your child's Duke Hospital and Clinic charges for as long as your child is in this study. These tests and studies are not a part of routine care, and people who are not part of the study do not usually have them performed. Please ask Dr. Smith if you and your child would like to know more about which tests and studies are being done solely for research purposes.

The study sponsor, CDC, has agreed to pay for services and procedures that are done solely for research purposes. Please talk with the Principal Investigator (Dr. Michael Smith) or study team about the specific services and procedures that the sponsor will pay for, and the ones for which you or your insurance will be responsible.

We will monitor your child's DUHS patient care charges to make sure that costs are directed appropriately. If you have any questions or concerns about appropriate billing, contact your study team coordinator so that he/she can help find a resolution.

#### WHAT ABOUT COMPENSATION?

All study participants will be compensated \$50 (to cover costs associated with parking, gas, and time) after completing each clinic visit, \$25 for each completed memory aid, and \$25 for each phone/telehealth visit. You will be paid for your child's participation in this study for the visits and activities completed.

Payment will be given only for study activities that are completed, for a maximum of \$175.

#### WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that your child is injured as a result of your child's participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your child's Duke physicians to provide monetary compensation or free medical care to your child in the event of a study-related injury.

For questions about the study or research-related injury, contact Dr. Michael Smith at 919-684-6335 during regular business hours and at (502) 235-4465 after hours and on weekends and holidays.

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW MY CHILD FROM THE STUDY?

You may choose not to allow your child to be in the study, or, if you agree to allow your child to be in the study, you may withdraw your child from the study at any time. If you withdraw your child from the study, no new data about your child will be collected for study purposes unless the data concern an adverse event (a bad effect) related to the study. If such an adverse event occurs, we may need to review your child's entire medical record. All data that have already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor (CDC).





Your decision to not allow your child to participate or to withdraw your child from the study will not involve any penalty or loss of benefits to which your child is entitled, and will not affect your child's access to health care at Duke.

If you decide to withdraw your child from the study, we ask that you contact Dr. Smith to let him know:

Dr. Michael Smith Box 102346 DUMC 315 Trent Drive Durham, NC 27710 michael.j.smith@duke.edu (919) 684-6335

The study doctor or sponsor may withdraw your child from this study for any reason at any time even without your consent. This could occur, for example, if the study doctor decides that it is in your child's best interest.

A description of this study will be available on <a href="https://clinicaltrials.gov/">https://clinicaltrials.gov/</a>. This website will not include information that can identify your child. At most, the website will include a summary of the results. You can search this website at any time.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you or your child have problems, concerns, questions or suggestions about the research, contact Dr. Smith at (919) 684-6335 during regular business hours and at (502) 235-4465 after hours and on weekends and holidays.

For questions about your child's rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.



Consent to Participate in a Research Study A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety of Simultaneous Vaccination with mRNA COVID-19 Vaccine and Other Vaccines in Young Children Aged 6 Months to <5 years.

# STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to allow my child to be in this study, with the understanding that I may withdraw my child at any time. I have been told that I will be given a signed and dated copy of this consent form.

| Signature of Parent/Guardian Date | Date | Time |
|---------------------------------------|------|------|
| Signature of Person Obtaining Consent | Date | Time |